CLINICAL TRIAL: NCT01719016
Title: Improvement Assessment of Coronary Flow Dysfunction Using Fundamental Fluid Dynamics
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Rupak K. Banerjee, Professor, University of Cincinnati
Other Study IDs: 10-05-05-02
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Reversible ischemia; microvascular dysfunction
MeSH Terms: conditions — Coronary Artery Disease | interventions — Adenosine; regadenoson

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Cardiac PET, Coronary catheterization: Cardiac PET scan:
  1. Injection of N-13 Ammonia radionuclide. 2 doses of 10 milliCuries and 20 milliCuries each.
  2. Injection of Lexiscan.
  Coronary catheterization:
  1. Pressure and flow readings using Combowire
  2. Injection of Adenosine.
  Interventions: Procedure: Cardiac PET, Coronary catheterization

INTERVENTIONS:
Procedure: Cardiac PET, Coronary catheterization — Patients would under go a Cardiac rest and stress PET scan and include the following drug administration:
  1. N-13 Ammonia radionuclide - Two doses, 10 mCi for rest, 20 mCi for stress
  2. Lexiscan - stress agent for PET scan
  Patients would also undergo Coronary catheterization including the following drug administration and device usage:
  1. Combowire to obtain pressure and flow readings on Combomap machine (Volcano Therapeutics, CA).
  2. Adenosine - stress agent during catheterization, 140 ug/Kg/min
  Other Names: Volcano therapeutics; Combomap machine; Adenosine; Lexiscan; N-13 Ammonia

SUMMARY:
Diagnosis of relative contributions of large artery blockages and microvascular blockages is very much needed in the treatment of coronary artery disease. In order to achieve this, two novel parameters, pressure drop coefficient (CDP), which combines flow and pressure readings and Lesion flow coefficient (LFC), which combines anatomical details of the lesion with pressure and flow readings, are being investigated.

DETAILED DESCRIPTION:
Diagnosis of relative contributions of large artery blockages and microvascular blockages is very much needed in the treatment of coronary artery disease. In order to achieve this, two novel parameters, pressure drop coefficient (CDP), which combines flow and pressure readings and Lesion flow coefficient (LFC), which combines anatomical details of the lesion with pressure and flow readings, are being investigated. The diagnostic parameters will be correlated with Coronary Flow Reserve (CFR)values obtained using Positron Emission Tomography (PET) imaging. They will also be correlated with Fractional Flow Reserve (FFR).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above
* Patients referred to a stress test by a Cardiologist
* Acute Chest pain, as per patient input.
* Risk Assessment with prior test results and/or previous history of known chronic stable CAD.
* Borderline or discordant stress testing where obstructive CAD remains a concern.
* New or worsening symptoms- Abnormal coronary angiography or abnormal prior stress imaging study.
* Coronary stenosis or anatomic abnormality of uncertain significance.
* In absence of reliable diagnostic information from another imaging modality.

Exclusion Criteria:

* Left ventricular ejection fraction less the 25% determined by gated SPECT imaging
* Non-dialysis dependent chronic kidney disease with baseline serum creatinine greater than 2.5 gm/dL.
* History of type II heparin-induced thrombocytopenia.
* Significant co-morbid condition that is medically unstable and would make coronary angiography prohibitive or contraindicated.
* Pregnant women.
* Incapacitated for Consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chest pain and suspected ischemia that needs to be assessed by a stress test
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-08; Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of relative contributions of large artery disease and microvascular disease | 2 years
  Correlation Coronary Flow Reserve (CFR) from Positron Emission Tomography (PET)imaging with diagnostic parameters, Pressure Drop Coefficient (CDP) and Lesion Flow Coefficient (LFC).

SECONDARY OUTCOMES:
Quantification of relative contributions of large artery disease and microvascular disease | 2 years
  Correlation of CDP and LFC with invasively measured Fractional Flow Reserve (FFR) values.

CONTACTS AND LOCATIONS:
Overall Officials: Rupak K Banerjee, PhD, Principal Investigator — University of Cincinnati , CVAMC; Mohamed Effat, MD, Principal Investigator — Univesity of Cincinnati, University Hospital; Imran Arif, MD, Principal Investigator — University of Cincinnati and University Hospital; Hanan Kerr, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Cincinnati Veteran Affairs Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Banerjee RK, Ramadurai S, Manegaonkar SM, Rao MB, Rakkimuthu S, Effat MA. Comparison Between 5- and 1-Year Outcomes Using Cutoff Values of Pressure Drop Coefficient and Fractional Flow Reserve for Diagnosing Coronary Artery Diseases. Front Physiol. 2021 Jul 14;12:689517. doi: 10.3389/fphys.2021.689517. eCollection 2021. PMID 34335296